CLINICAL TRIAL: NCT06537037
Title: Exploring the Association of Imaging and Tumor Microenvironment in Urologic Cancer Using Radiogenomic Approach（Radiogenomics-Urinary）
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: S187
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Urologic Cancer
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is the prospective, observational cohort study (Radiogenomics-Urinary), which aims to explore the relationship between the imaging information of urologic cancer patients, tumor microenvironment and the prognosis of urologic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated for urologic cancer in Wuhan Union Hospital from August 2024 to August 2027;
2. Aged > 18 years old;
3. At least one CT scan or MRI scan before treatment;
4. Tissue biopsy pathological examination confirmed the diagnosis of the above tumors.

Exclusion criteria：

1. Poor image quality;
2. Incomplete clinical data or loss of follow-up;
3. Presence of another primary malignancy other than urologic cancer;
4. Unclear pathological diagnosis。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for urologic cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Correlation analysis of sequencing results and body composition | 0.5 year
  Conducting correlation analysis between body composition and results of multi-omics sequencing.
Correlation analysis of sequencing results and tumor radiomic features | 0.5 year
  Conducting correlation analysis between radiomic features and results of multi-omics sequencing.

SECONDARY OUTCOMES:
Constructing tumor microenvironment prediction model | 2 years
  Constructing radiomic model to predict tumor microenvironment. The indicator is the area under the curve (AUC) of the prediction model
Constructing a multi-dimensional prognostic prediction model | 3 years
  A high-dimensional model was constructed to predict the prognosis of patients through multi-omics sequencing data, body composition, and tumor radiomic features. The indicator is the area under the curve (AUC) of the prediction model.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China